CLINICAL TRIAL: NCT02651805
Title: Mechanical Insufflator-exsufflator to Manage Respiratory Secretion in Patients in Palliative Care - A Feasibility Study
Brief Title: Mechanical Insufflator-exsufflator to Control Mucus Hypersecretion in Patients in Palliative Care - A Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Hospital Estadual Américo Brasiliense (Unknown); Philips Respironics (Industry)
Responsible Party: Principal Investigator, Juliano Ferreira Arcuri, PhD Student, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MIE-Palliative
Record Dates: First submitted 2015-12-16; First posted 2016-01-11 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Palliative Care; Mucus Hypersecretion
Keywords: Palliative Care; Respiratory Secretion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mechanical Insufflation-Exsufflation Group (Experimental): Patients will receive usual care except suctioning or cough augmentation techniques+Mechanical Insufflation-Exsufflation
  Interventions: Device: Mechanical Insufflation-Exsufflation
- Usual Care Group (Active Comparator): Patients will receive the usual care provided by the hospital, all interventions to control respiratory secretion will be verified in patient chart
  Interventions: Device: Mechanical Insufflation-Exsufflation; Other: Usual Care

INTERVENTIONS:
Device: Mechanical Insufflation-Exsufflation — Mechanical Insufflator-Exsufflator (MI-E): 6 assisted cough with expiratory pressure of -40cmH2O and inspiratory pressure defined by the therapist as the maximum pressure defined as comfortable; inspiratory time 3s and expiratory time 4s, using a manual cycle. Patients will be instructed to cough during exsufflation phase, with exception of Chronic obstructive pulmonary disease patients which will be instructed to exhale slowly. An oral-nasal mask will be used as interface, but in patients with tracheotomy, the device will be connected to it. A trained physiotherapist will conduct the therapy. During the night and weekends, patients will not start this therapy, however, if they have already started the therapy in MI-E group, or if they have already finished the period of follow-up they will be able to request this therapy, which will be provided by hospital staff . The equipment (Cough Assist®, Respironics, Phillips), will be available in the ward for the interventions.
  Other Names: Cough Assist (Philips Respironics)
Other: Usual Care — The patients will receive the treatment according to the hospital protocol to deal with hypersecretive patients (suctioning that can be preceded by respiratory physiotherapy and nebulisation). A trained member of the nurse staff or a physiotherapist will be responsible for providing the therapy. A member of the research team will collect in the patients' records all the therapies provided by the staff to control hypersecretions.
  Arms: Usual Care Group

SUMMARY:
Patients with advanced chronic diseases may suffer with respiratory secretion and available therapies to control this condition are uncomfortable or little effective in palliative care patients. Therefore, alternative therapies should be tested, assessing clinically relevant outcomes in palliative care, such as comfort during therapy and the number of interventions required in a day. Mechanical Insufflation-Exsufflation is an option that presents advantages, since it can be used in patients with minimum cooperation and is non-invasive, which may lead to higher comfort during therapy.

The aim of the study is to verify the feasibility of a clinical trial comparing the effects of Mechanical Insufflation-Exsufflation with usual care in hospitalized palliative care patients that are suffering with respiratory secretion. Patients allocation will follow a "fast-track allocation design", in which included patients will be randomized in two groups:

1. Receive Mechanical Insufflation-Exsufflation therapy in the moment that is assigned to this group;
2. will receive 24h of usual care and after that will be allowed to choose between usual care or Mechanical Insufflation-Exsufflation Therapy.

The assessments will be: Time from the first intervention until the need of a following intervention, discomfort due therapy, discomfort due respiratory secretion, palliative outcome scale, number of adverse events and number of interventions during 24h period. The primary outcome is to verify the feasibility of developing a future larger clinical trial to assess the effects of the use of Mechanical Insufflation-Exsufflation to control respiratory secretions in patients in palliative care.

DETAILED DESCRIPTION:
Investigators will conduct a feasibility study for a future fast track randomized trial, which will be carried out in the Américo Brasiliense State Hospital and conducted by the Spirometry and Respiratory Physiotherapy Laboratory from the Federal University of São Carlos, Brazil.

The concept of feasibility is defined as "capable of being done or carried out" and studies which aim is to verify the feasibility intends to verify if a larger clinical trial would have a acceptable probability of success in proving the efficacy of an intervention 24. The importance of feasibility studies has been discussed since health research resources are frequently wasted in large clinical trials with interventions with small impact, studies with insufficient power, or even using measures and outcomes that do not reflect the expected changes caused by the interventions. Furthermore, these studies are essential when dealing with populations that usually lead to an increased chance of losing the follow-up or a high number of missing data, such as palliative care.

Both groups will receive the therapy with the mechanical insufflators-exsufflator, however, the Mechanical insufflation-exsufflation group will receive it as in a fast track way, while the usual care, will receive the usual care for more 24 hours, and then they will receive one session of Mechanical Insufflation-Exsufflation. After this 24 hours period, the patients will be asked what therapy they would like to receive each time they need help to deal with hypersecretion until the end of the hospitalization, or until the physician responsible for the patient consider the hypersecretion was controlled.

The allocation through fast track has been used due to ethical reasons, in order to maintain the randomized and controlled aspects of the research, and yet provide the opportunity to all patients to be benefited of the new intervention before the end of the study. Furthermore, an increase in the acceptability and retention of the participants is expected, since they are going to receive the new therapy in some moment of the study, which may be during or after the follow-up 28. The cross-over design was not chosen, since the wash-out period necessary to this model of study might lead to a period without treatment for vulnerable patients, with expected short life time.

Usual Care The patients will receive the treatment according to the hospital protocol to deal with hypersecretive patients (suctioning that can be preceded by respiratory physiotherapy and nebulisation). A trained member of the nurse staff or a physiotherapist will be responsible for providing the therapy. A member of the research team will collect in the patients' records all the therapies provided by the staff to control hypersecretions.

Mechanical Insufflation-Exsufflation The settings used in the Mechanical Insufflator-Exsufflator will be the same of a previous study, where were used: six assisted cough cycles with pressures of 40 to -40cmH2O; the inspiratory time of 3s; the expiratory time 4s and a pause between cycles of 4s. The patients will be instructed to cough alongside the exsufflation phase, with exception of Chronic Obstructive Pulmonary Disease patients which will be instructed to exhale slowly. An oral-nasal mask will be used as interface, but in patients with tracheotomy, the device will be connected to it.

ELIGIBILITY:
Inclusion Criteria:

* Prognosis:

  * Less than one year assessed by the responsible physician, with a negative answer of the to the "surprise question" - Would you be surprised if this patient died in the following year?
  * Higher than 3 months, assessed by the same physician
* Patients with problems to deal with secretions, which could be one or both of the following problems:

  * Hypersecretion
  * Cough inefficiency (peak cough flow <250L/min)
* Karnofsky Performance Status Scale higher or equal to 30%;
* Ability to give written informed consent or presence of a person who is responsable for the patient

Exclusion Criteria:

* Patients with conditions considered as contra-indication for the use of Mechanical Insufflator-Exsufflator:

  * Bullous emphysema history
  * Known susceptibility for pneumothorax or pneumo-mediastinum
  * Known to have had any recent barotrauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07-30 (Estimated); Study Completion 2017-07-30 (Estimated)

PRIMARY OUTCOMES:
Study Feasibility assessed by verifying the recruitment rates, acceptability of the patients and hospital | Through the completion of the study, up to one year
  The feasibility of the study will be the primary outcome, and it will be assessed by verifying the recruitment rates, acceptability of the patients and hospital, and if the assessments were suitable to the study

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Assessed in the period between the start of the intervention until 30min after the end of the intervention
  Assessed by the number of times an event with change in physiological parameters occurred during the intervention (Heart Rate>150bpm or <50bpm; Systolic Blood Pressure>200mmHg or <80mmHg; decrease of 5% or higher in the pulse oxymetry; hemoptysis).
Effect size of Palliative Outcome Scale | Immediately after the inclusion and in the final assessment (24 hours after the inclusion).
  This is a quality of life multidimensional scale in patients in palliative care. With this scale, we intend to see the effects of the therapy over the general perceived health of the patients.
Effect size of discomfort due to the hypersecretion | Immediately before the first intervention and ten minutes after the first intervention.
  Assessed using a numeric scale (0-10). This assessment will be conducted in order to evaluate how much the hypersecretion bothers the patient, and if the therapy is capable of changing this perception of discomfort.
Effect size of discomfort due to the therapy | Ten minutes after the first intervention
  Assessed using a numeric scale (0-10), this assessment will provide information to the decision of the viability the therapy in palliative care, since uncomfortable therapies are often discouraged since usually they may not cure the cause of the problem.
Effect size of time until the next intervention | In the end of the 24 hours period.
  The moment immediately after the first intervention until the time a new intervention is required. It will be verified in the patient's records. The therapies to control hypersecretions may lead to discomfort due to the stimulation of the cough and the change in the respiratory pattern, a therapy with a more lasting effect may be preferable, since it can provide a longer period without the discomfort of another intervention.
Effect size of number of interventions during 24 hours | In the end of the 24 hours period
  The number of interventions will be verified in the patient's records. Therapies that may lead to a lasting effect, can be performed less times during a day, this reflects in a longer period of comfort, and smaller health expenses.

OTHER OUTCOMES:
Percentage of patients using pharmacological agents to control respiratory secretions | In the completion of the study, an average of one year
  Patient's chart will be revised to verify the percentage of patients that received pharmacological interventions to control respiratory secretions, prescribed by the hospital team.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Estadual Américo Brasiliense, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bach JR. Mechanical insufflation-exsufflation. Comparison of peak expiratory flows with manually assisted and unassisted coughing techniques. Chest. 1993 Nov;104(5):1553-62. doi: 10.1378/chest.104.5.1553. PMID 8222823
- [Background] Bach JR. Amyotrophic lateral sclerosis: prolongation of life by noninvasive respiratory AIDS. Chest. 2002 Jul;122(1):92-8. doi: 10.1378/chest.122.1.92. PMID 12114343